CLINICAL TRIAL: NCT00057304
Title: A Phase II Randomized, Double-Blind, Dose-Ranging Study to Determine the Efficacy, Safety, Tolerability & Pharmacokinetics of RO 205-2349 in Patients With Type 2 Diabetes Mellitus
Brief Title: Study to Determine the Efficacy, Safety, Tolerability & Pharmacokinetics of RO 205-2349 in Patients With Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM17151
Record Dates: First submitted 2003-03-31; First posted 2003-04-01 (Estimated); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus | interventions — BM 13.1258

STUDY DESIGN:
Intervention Model Description: All potential participants entered the placebo run-in phase. At the end of the placebo run-in phase, eligible participants who met the final inclusion/exclusion criteria were randomized to the double-blind treatment period.
  treatment
Who Masked: Participant, Investigator

ARMS (2):
- RO 205-2349 2 mg QD (Experimental): RO 205-2349 2 mg was taken once daily (QD) for 16 weeks during the double-blind treatment period.
  Interventions: Drug: RO 205-2349
- RO 205-2349 5 mg QD (Experimental): RO 205-2349 5 mg was taken once daily (QD) for 16 weeks during the double-blind treatment period.
  Interventions: Drug: RO 205-2349

INTERVENTIONS:
Drug: RO 205-2349
  Other Names: Edaglitazone

SUMMARY:
The objective of the study is to determine the dose(s) of Ro 205-2349 which, when compared to placebo, are efficacious, safe and tolerable in improving glycemic control in patients with type 2 diabetes. Doses of 2 to 5 mg/day will be studied.

ELIGIBILITY:
Inclusion Criteria:

* Age 35 to 75
* Type 2 diabetes for longer than 3 months
* HbA1c (glycosylated hemoglobin A1c) greater than 7.0% at screening
* FPG (fasting plasma glucose) greater than 126 mg/dL at screening
* BMI (body mass index) less than 40 kg/square meter

Exclusion Criteria:

* Type I diabetes
* Type 2 diabetes patients currently treated with insulin
* Type 2 diabetes patients currently or previously treated with Actos, Avandia or Rezulin
* FPG (fasting plasma glucose) greater than 270 mg/dL at baseline
* Impaired liver or kidney function
* Triglycerides greater than 600 mg/dL
* Uncontrolled hypertension
* Pregnant or lactating women
* Women not using adequate contraception

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 190 (Actual)
Dates: Start 2003-06 (Actual); Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (38):
- United States (12):
  - Hollywood, Florida
  - Durham, North Carolina
  - Morrisville, North Carolina
  - Portland, Oregon
  - Camp Hill, Pennsylvania
  - Greer, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Houston, Texas
  - Midland, Texas
  - Lebanon, Virginia
  - Virginia Beach, Virginia
- Bulgaria (3):
  - Pleven
  - Plovdiv
  - Sofia
- Estonia (3):
  - Tallinn
  - Tartu
  - Võru
- Mexico (7):
  - Chihuahua, Chih.
  - Guadalajara
  - Guadalajara, JAL.
  - Mexico City
  - Mérida
  - Monterrey
  - Pachuca, Hidalgo
- Panama City, Panama
- Ponce, Puerto Rico
- Romania (8):
  - Arad
  - Brasov
  - Bucharest
  - Craiova
  - Galati
  - Ploieşti
  - Târgovişte
  - Târgu Mureş
- Meyrin, Switzerland
- United Kingdom (2):
  - Bracknell
  - Nottingham